CLINICAL TRIAL: NCT05288322
Title: The Effectiveness of Mostafa Maged Maneuveur to Prevent and Control Post-partum Haemorrhage During Normal Vaginal Delivery
Brief Title: Mostafa Maged Maneuveur to Prevent and Control Post-partum Haemorrhage During Normal Vaginal Delivery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fayoum University (Other)
Responsible Party: Principal Investigator, Mostafa Maged Ali, Principal investigator, Fayoum University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: R218
Record Dates: First submitted 2022-03-08; First posted 2022-03-21 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: Post Partum Hemorrhage
Keywords: Mostafa Maged maneuver; Atony; normal delivery; postpartum bleeding
MeSH Terms: conditions — Postpartum Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mostafa Maged maneuver to prevent and control post-partum haemorrhage (Experimental): all pregnant females ( primigravida and multi-gravida ) . this study includes forty pregnant females with normal vaginal delivery .this study includes pregnant females Inclusion criteria :-
  1. All pregnant patients
  2. Age is between (18) to (40) years old
  The Mostafa Maged maneuveur has been applied to those all female patients to prevent or control post-partum bleeding in normal delivery .
  Interventions: Procedure: Mostafa Maged maneuver

INTERVENTIONS:
Procedure: Mostafa Maged maneuver — The Mostafa Maged maneuveur has been applied to those all female patients to prevent or control post-partum bleeding in normal delivery . The Mostafa Maged technique is applied by :- (Description of the new Mostafa Maged technique) :-
  1. First , placing our right hand to the posterior fornix of vaginal canal trying to cuddle the lower part of uterus compressing the anterior and posterior walls of the uterus .
  2. Second , placing our left hand over the fundus of the uterus and the posterior wall of uterus from the abdominal part.
  3. Third , by our two hands , trying to grasp the whole uterus by our two hands abdominally and vaginally against the symphysis pubis as if the uterus is cuddling the symphysis pubis bone and in this way , we try to get the anterior and posterior walls against each other and reducing the intra-cavitary space so we prevent the expansion of the uterus .

SUMMARY:
PPH is commonly defined as blood loss exceeding 1000 milliliters after vaginal birth or cesarean section.1 PPH is often classified as primary/immediate/early (occurring within 24 hours of birth) or secondary/delayed/late (occurring from more than 24 hours postbirth to up to 12 weeks postpartum)..

Atonic post-partum haemorrhage is one of the most challenging complications of normal delivery process . There are many maneuveurs applied to the atonic uterus for controlling the blood loss and conserving the uterus from hysterectomy process . There are pharmacological and surgical methods to control the bleeding . In this study , Mostafa Maged technique is to prevent and control post-partum bleeding during vaginal delivery . It is so simple and not-costly method .

DETAILED DESCRIPTION:
In this study , Mostafa Maged technique to prevent and control post-partum bleeding during vaginal delivery . It is so simple and not-costly method . Mostafa Maged maneuveur has been applied to those all female patients to prevent or control post-partum bleeding in normal delivery . Mostafa Maged technique is applied by :- (Description of the Mostafa Maged technique) :-

1. First , placing the right hand to the posterior fornix of vaginal canal trying to cuddle the lower part of uterus compressing the anterior and posterior walls of the uterus .
2. Second , placing the left hand over the fundus of the uterus and the posterior wall of uterus from the abdominal part of the pregnant mother ( the side of the abdominal skin ) .
3. Third , by the two hands , trying to grasp the whole uterus by the two hands abdominally and vaginally against the symphysis pubis as if the uterus is cuddling the symphysis pubis bone and in this way , getting the anterior and posterior walls of the uterus against each other compressed is achieved and reducing the intra-cavitary space so prevention of the expansion of the uterus is applied .

ELIGIBILITY:
Inclusion Criteria:

* pregnant females Inclusion criteria :-

  1. All pregnant patients
  2. Age is between (18) to (40) years old

Exclusion Criteria:

1. Smokers
2. Morbid obese
3. Medical history of blood diseases and collagen diseases

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2022-04-10 (Actual); Primary Completion 2022-05-20 (Actual); Study Completion 2022-05-20 (Actual)

PRIMARY OUTCOMES:
post-partum bleeding | six hours post-delivery
  prevention and treatment of post-partum bleeding in normal vaginal delivery by estimating the number of pads used during normal delivery to see amount of blood loss and to estimate the blood loss visually roughly as well

CONTACTS AND LOCATIONS:
Locations (1):
- Fayoum general hospital and Fayoum university, Al Fayyum, Egypt

IPD SHARING:
Plan to Share IPD: No